CLINICAL TRIAL: NCT05227586
Title: Adjunctive Right Atrial Ablation for Persistent Atrial Fibrillation With Right Atrial Enlargement
Status: Completed | Type: Observational
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Xu Liu, Professor, deputy director of cardiology department of Shanghai Chest Hospita, Shanghai Chest Hospital
Other Study IDs: RAAFDA
Record Dates: First submitted 2022-01-26; First posted 2022-02-07 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Persistent Atrial Fibrillation; Right Atrial Enlargement
Keywords: Atrial fibrillation; Right atrium
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LA + RA ablation: Patients with persistent atrial fibrillation and right atrial enlargement received adjunctive right atrial ablation when left atrial ablation did not terminate atrial fibrillation.
  Interventions: Procedure: Circumferential pulmonary vein isolation + linear ablation + bi-atrial mapping + left atrial driver ablation + right atrial driver ablation
- LA ablation only: Patients with persistent atrial fibrillation and right atrial enlargement received left atrial ablation only
  Interventions: Procedure: Circumferential pulmonary vein isolation + linear ablation + bi-atrial mapping + left atrial driver ablation

INTERVENTIONS:
Procedure: Circumferential pulmonary vein isolation + linear ablation + bi-atrial mapping + left atrial driver ablation — Patients receive circumferential pulmonary vein isolation and linear ablation (ablation of a roof line and a mitral isthmus line) combined with bi-atrial mapping and left atrial driver ablation.
  Groups: LA ablation only
Procedure: Circumferential pulmonary vein isolation + linear ablation + bi-atrial mapping + left atrial driver ablation + right atrial driver ablation — Patients receive circumferential pulmonary vein isolation and linear ablation (ablation of a roof line and a mitral isthmus line) combined with bi-atrial mapping , left atrial driver ablation and right atrial driver ablation.
  Groups: LA + RA ablation

SUMMARY:
This is retrospective cohort study testing whether patients with persistent atrial fibrillation and right atrial enlargement may benefit from adjunctive right atrial ablation.

DETAILED DESCRIPTION:
This is retrospective cohort study testing whether patients with persistent atrial fibrillation and right atrial enlargement may benefit from adjunctive RA ablation.

We enrolled 65 patients with persistent atrial fibrillation and right atrial enlargement received adjunctive right atrial ablation. These patients were 1:2 match with 130 patients received left atrial ablation only. Atrial fibrillation recurrence rate and other paremeters were analyzed to evaluate the efficacy of adjunctive right atrial ablation in this subset of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 80 years old;
2. Persistent AF with right atrial enlargement;
3. Nonresponse or intolerance to ≥1 antiarrhythmic drug.

Exclusion Criteria:

1. History of catheter ablation;
2. valvular heart disease;
3. hypertrophic cardiomyopathy or dilated cardiomyopathy;
4. Without follow-up data

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population enrolled were patients with persistent atrial fibrillation and right atrial enlargement received catheter ablation for the first time in our institution.
  Patients with a history of catheter ablation, valvular heart disease, hypertrophic or dilated cardiomyopathy and unavailable of follow-up data were excluded
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
atrial fibrillation (AF) recurrence rate | at 12 months post procedure
  AF recurrence is defined as presence of documented AF episodes of 30 seconds or longer duration

SECONDARY OUTCOMES:
atrial fibrillation (AF)/atrial flutter (AFL)/atrial tachycardia (AT) recurrence rate | at 12 months post procedure
  AF/AFL/AT recurrence is defined as presence of documented AF/AFL/AT episodes of 30 seconds or longer duration

CONTACTS AND LOCATIONS:
Locations (1):
- Mu Qin, Shanghai, China